CLINICAL TRIAL: NCT06511583
Title: FBS-ASaP: Fibrobronchoscopy in ASpiration Pneumonia in the Emergency Department
Acronym: FBS-ASaP
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Principal Investigator, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: CEAVC 22814
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Aspiration Pneumonia; Bronchoscopy
Keywords: Aspiration pneumonia; Bronchoscopy; toilette; interventional pulmunology; respiratory failure; pneumonia; bacterial pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration; Respiratory Insufficiency; Pneumonia; Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laryngotracheal Aspiration Procedure Using a Probe in the Emergency Department: Patients with aspiration pneumonia. For laryngotracheal aspiration using a blind probe, the patient will be positioned in a seated or semi-seated position; if this is not possible, the aspiration will be performed in a supine position. A soft, sterile catheter connected to the suction apparatus will be inserted into one nostril while keeping the patient's head tilted back. When the tip of the catheter reaches the back of the pharynx, the patient will need to breathe to facilitate the insertion and allow the catheter to advance into the larynx and trachea. At this point, using negative suction pressure for a maximum of 3-5 seconds, the secretions will be aspirated. The aspiration will be repeated multiple times in cycles of 3-5 seconds.
  Interventions: Procedure: Laryngotracheal Aspiration Procedure Using a Probe in the Emergency Department
- Aspiration Using Fibrobronchoscopy in the Emergency Department: Patients with aspiration pneumonia. The bronchoscope will be gently inserted through the patient's nostril or mouth, advancing carefully through the pharynx and larynx into the trachea and bronchi.
  The physician will visually inspect the airways through the bronchoscope. Using the bronchoscope's suction channel, secretions will be aspirated from the trachea and bronchi.
  Suctioning will be performed intermittently to avoid hypoxia, with each suctioning cycle lasting no more than 3-5 seconds.
  The procedure may be repeated as necessary to ensure thorough aspiration of secretions.
  Interventions: Procedure: Aspiration Procedure Using Fibrobronchoscopy in the Emergency Department

INTERVENTIONS:
Procedure: Laryngotracheal Aspiration Procedure Using a Probe in the Emergency Department — For laryngotracheal aspiration using a blind probe, the patient will be positioned in a seated or semi-seated position; if this is not possible, the aspiration will be performed in a supine position. A soft, sterile catheter connected to the suction apparatus will be inserted into one nostril while keeping the patient's head tilted back. When the tip of the catheter reaches the back of the pharynx, the patient will need to breathe to facilitate the insertion and allow the catheter to advance into the larynx and trachea. At this point, using negative suction pressure for a maximum of 3-5 seconds, the secretions will be aspirated. The aspiration will be repeated multiple times in cycles of 3-5 seconds.
  Groups: Laryngotracheal Aspiration Procedure Using a Probe in the Emergency Department
Procedure: Aspiration Procedure Using Fibrobronchoscopy in the Emergency Department — Equipment Setup:
  A sterile bronchoscope will be connected to the suction apparatus.
  Procedure:
  The bronchoscope will be gently inserted through the patient's nostril or mouth, advancing carefully through the pharynx and larynx into the trachea and bronchi.
  The physician will visually inspect the airways through the bronchoscope. Using the bronchoscope's suction channel, secretions will be aspirated from the trachea and bronchi.
  Suctioning will be performed intermittently to avoid hypoxia, with each suctioning cycle lasting no more than 3-5 seconds.
  The procedure may be repeated as necessary to ensure thorough aspiration of secretions.
  Groups: Aspiration Using Fibrobronchoscopy in the Emergency Department

SUMMARY:
Non-Profit Prospective Observational Pilot Study

The study will have an overall duration of 3 years, with patient enrollment starting after ethical committee approval.

In this study, all patients with a diagnosis of aspiration pneumonia who require aspiration of secretions or ingesta in the Emergency Department will be considered. A registry will be created with the patients' data, noting the type of procedure performed: laryngotracheal aspiration with a probe or with fibrobronchoscopy.

This observational registry pilot study aims to evaluate the utility and adverse events related to the use of aspiration via videobronchoscopy performed in the Emergency Department and to compare the clinical outcomes of patients undergoing bronchoscopy with those treated only with blind laryngotracheal aspiration using a probe.

ELIGIBILITY:
Inclusion Criteria:

All adult patients who access the Emergency Department with a diagnosis of aspiration pneumonia and for whom the referring physician determines the need for aspiration of secretions or ingesta. Patients must have at least one of the following criteria

* Radiological evidence of pneumonia (Chest X-ray/CT scan/Chest ultrasound)
* Clinical diagnosis of aspiration pneumonia
* Presence of secretions in the upper airways
* Respiratory distress in a dysphagic patient
* Need for oxygen therapy or need to increase FiO2 in patients already on home oxygen therapy

Exclusion Criteria:

* Lack of consent
* Age < 18 years
* Pregnancy
* Hemorrhagic diathesis
* Malignant cardiac arrhythmias (VT, AV block excluding first-degree AV block)
* Severe airway obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on patients with a diagnosis of aspiration pneumonia who, based on the judgment of the attending physician, require aspiration of secretions or ingesta in the emergency department using a probe and/or a fiberscope. Enrollment in the study will be determined by the Emergency Department physician in charge of the patient.
  Estimated number of patients to be enrolled: 100.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay in days | up to 3 months
  Length of hospital stay in days
Mortality rate within 30 days from the time of admission to the Emergency Department | 30 days from admission to the ed
  Mortality rate within 30 days from the time of admission to the Emergency Department

SECONDARY OUTCOMES:
Respiratory parameters before and after the procedure | on the admission and 30 minutes after the procedure
  (SpO2, FiO2)before and after the procedure
Rate of patient treated with Non invase ventilation and with orotracheal intubation | on the admission and 30 minutes after the procedure
  Oxygen therapy devices before and after the procedure
Rate of admission in Intensive care unit and High dependency unit | immediately after the procedure
  Hospitalization setting
Procedure-related complications | perioperatively/periprocedurally
  Procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Pelagatti, dr, Principal Investigator — University of Florence
Locations (1):
- AOU Careggi, Florence, Tuscany/Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided